CLINICAL TRIAL: NCT06088862
Title: A Randomized Study to Evaluate Harm Reduction Products as a Second Line Intervention for Adult Smokers Who Do Not Quit With Nicotine Replacement Therapy (NRT)
Brief Title: Evaluate Harm Reduction Products as a Second Line Intervention for Adult Smokers Who Do Not Quit With NRT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: BIDI product received a market denial letter from the FDA
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adaptive
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Harm Reduction
MeSH Terms: conditions — Smoking Cessation; Harm Reduction | interventions — Nicotine; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group I - NRT Responder (Experimental): Participants that were successful in quitting smoking using NRT in the first four weeks of the study will have the option of remaining on their current NRT or switching to one of the other two options for the next five weeks.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product
- Group IIa NRT Non-Responder - Pouch Preferrers (Experimental): Participants that were unsuccessful in quitting smoking using NRT in the first four weeks and reported a preference to try a nicotine pouch. Randomized to be switched to nicotine pouch for the next five weeks.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product; Other: on!
- Group IIb NRT Non-Responder - Pouch Preferrers Control (Experimental): Participants that were unsuccessful in quitting smoking using NRT in the first four weeks and reported a preference to try a nicotine pouch. Randomized to be remain on NRT for the next five weeks.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product
- Group IIIa NRT Non-Responder - ENDS Preferrers (Experimental): Participants that were unsuccessful in quitting smoking using NRT in the first four weeks and reported a preference to try ENDS. Randomized to be switched to ENDS for the next five weeks.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product; Other: BIDI e-cigarette
- Group IIIb NRT Non-Responder - ENDS Preferrers Control (Experimental): Participants that were unsuccessful in quitting smoking using NRT in the first four weeks and reported a preference to try ENDS. Randomized to be remain on NRT for the next five weeks.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product

INTERVENTIONS:
Drug: Nicoderm — 21mg nicotine patch daily; maximum usage 9 weeks
  Other Names: Nicotine Patch
Drug: Nicorette 4Mg Chewing Gum — 4mg Nicorette gum (flavors - cinnamon surge, fruit chill, and mint); as needed maximum usage 9 weeks
  Other Names: Nicotine gum
Drug: Nicorette Lozenge Product — 4mg Nicorette mint lozenge; as needed maximum usage 9 weeks
  Other Names: Nicotine lozenge
Other: BIDI e-cigarette — BIDI e-cigarette (flavors - Classic, Arctic, and Solar); as needed for maximum of 5 weeks
  Arms: Group IIIa NRT Non-Responder - ENDS Preferrers
Other: on! — 4mg on! Nicotine Pouch (flavors - Berry, Mint, and Original); as needed for maximum usage 5 weeks
  Other Names: Nicotine pouch
  Arms: Group IIa NRT Non-Responder - Pouch Preferrers

SUMMARY:
This study will determine whether a range of products along the reduced-risk continuum can reduce smoke exposure for individuals who fail to quit smoking using current medically approved nicotine replacement therapy (NRT) products. The strategy will be to offer 325 smokers four weeks of NRT of their choice (gum, lozenge, or nicotine patch) and assess them for quit-smoking status at the end of the period. Seven-day point abstinence will be used to determine responder status at the end of the four-week period (CO of <6 ppm at both CO collection points during that seven-day period and self-report of no smoking during that seven-day period). Those who have not quit, and who therefore have a very low chance of later success (a consistent finding in prior studies and to be verified in the proposed study), will be randomly assigned to either receive a potential "rescue" product (nicotine pouch or ENDS (electronic nicotine delivery system), or remain on NRT (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the Informed Consent From (ICF) and is able to read and understand the information provided in the ICF.
2. Is 22 to 65 years of age (inclusive) at screening.
3. Smokes an average of at least 10 commercially available cigarettes per day and has done so for the last 12 months.
4. Expired air CO reading of at least 10 ppm as assessed at the screening session.
5. Interested in switching to an electronic cigarette or nicotine pouch.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Any participant who has a medical or physical condition that, in the opinion of the investigator (or designee), may adversely affect participant safety, the safety of others, or data validity.
2. Planned use of an FDA-approved smoking cessation product during the study, not provided as part of this protocol.
3. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
4. Taking psychoactive medications (e.g., antipsychotics, benzodiazepines, or mood stabilizers).
5. Frequent users (monthly) of smokeless tobacco (chewing tobacco, snuff), cigars (not cigarillos), pipes, hookahs or other non-commercially available combustible or heated tobacco products.
6. Use of nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
7. Pregnant or nursing (by self-report) or positive pregnancy test.
8. Heterosexually active participant of Childbearing Potential (not sterilized by tubal ligation, oophorectomy, hysterectomy, or other surgical methods, or post-menopausal) that do not agree to practice medically appropriate methods of birth control (or remain abstinent) during the course of the trial. Medically acceptable methods of birth control include: successful vasectomy of male partner, vaginal diaphragm with spermicide, intrauterine device, hormonal birth control (oral, injected, or implanted), condom with spermicide, or sponge with spermicide.
9. Participants who were enrolled in a clinical trial within 30 days of screening.
10. Enrollment numbers met (in sub-group or entire study).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in smoke exposure for NRT non-responders | After 10 weeks
  Change in expired air CO at week 10 compared to baseline

SECONDARY OUTCOMES:
Smoking abstinence rates for NRT non-responders | Week 7 - Week 10
  Complete smoking abstinence defined by a self-report of no cigarette smoking (not even a puff).
Smoking abstinence rates for NRT non-responders | Week 7 - Week 10
  Complete smoking abstinence defined by expired air CO<6 ppm.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No